CLINICAL TRIAL: NCT05838534
Title: Microbiome Comparison Profile of Normal Skin and Acne Vulgaris Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, SpKK - Head of Cosmetic Dermatology Division, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Organization: Indonesia University (Other)
Other Study IDs: SkinMicrobiomeComparison
Record Dates: First submitted 2023-04-05; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Acne Vulgaris
Keywords: Skin Microbiome; Normal Skin; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Skin
- Mild Acne Vulgaris
- Moderate Acne Vulgaris
- Severe Acne Vulgaris

SUMMARY:
The aim of this study is to compare the profile of the microbiome on normal skin and acne vulgaris patients. A cross sectional study with 144 samples, male or female between 18-40 years old, from January to May 2023.

DETAILED DESCRIPTION:
Recently, research on the role of the microbiome in the process of acne vulgaris has continued to grow. Seeing the important role of the microbiome in maintaining the balance of skin health, this study aims to compare the profile of the microbiome on normal skin and on acne vulgaris patients, in order to gain a deeper understanding the role of the microbiome in acne vulgaris and also to compare skin microbiome features in various degrees of acne vulgaris severity. This research is an observational study with a cross sectional design. Subject selected by consecutive sampling, with total 144 samples consists of males and females age 18-40.

There will be two visits in this research. The first visit, for screening patients with requests for informed consent, giving facial soap, screening for inclusion and exclusion criteria, screening for facial skin complaints and facial care habits, collecting data on patient demographics and medical history, physical examination, sebumeter examination to measure sebum levels on facial skin, and taking clinical photos for documentation. The second visit is collecting microbiome data which will be taking in 1 to 2 weeks after the first visit. Using swab method to take microbiome samples, after that, there will be DNA extraction, amplification and sequencing were carried out on the sample and the Shannon Index will be calculated. Then, the data will be tabulated and analyzed according to the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-40 years old
* Normal individuals who have not had acne vulgaris in the last 5 years and have never had moderate or severe acne vulgaris
* Patients with mild, moderate, or severe acne vulgaris who have acne vulgaris lesions that are representative of the grade and equally distributed in all facial regions (forehead, cheeks, and chin)
* Patients agree to participate in the study and sign informed consent

Exclusion Criteria:

* Pregnancy
* Diagnosed with other inflammatory or infectious diseases on the face
* Diagnosed with psoriasis or have atopic
* Diagnosed with primary or secondary immunodeficiency disease
* Patients with a history of laser therapy or facial dermabrasion within the past month
* Using oral or systemic antibiotics, anti-inflammatory, retinoids or hormone therapy in the last 1 month
* Using topical retinoid therapy, antibiotics, benzoyl peroxide, or other topical products in the last 2 weeks
* Acne conglobata

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male or female, 18-40 years old, normal skin, diagnosed with mild to severe acne
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-05-24 (Estimated)

PRIMARY OUTCOMES:
Comparison of skin microbiome features on normal and acne vulgaris skin | up to 16 weeks
  Using the swab method on facial skin for microbiome sampling, DNA extraction, amplification, and sequencing were carried out on the sample and the Shannon Index will be calculated. Then, the data will be tabulated and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Irma Bernadette Sitohang, MD, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (2):
- Indonesia (2):
  - Clinical Research Supporting Unit- Faculty of Medicine, University of Indonesia, Jakarta Pusat, DKI Jakarta
  - Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta

REFERENCES:
- [Derived] Manurung THP, Sitohang IBS, Agustin T. Staphylococcus caprae and Staphylococcus epidermidis define the skin microbiome among different grades of acne vulgaris. Arch Dermatol Res. 2024 Dec 30;317(1):156. doi: 10.1007/s00403-024-03581-1. PMID 39738874